CLINICAL TRIAL: NCT01878006
Title: OPRM1 A118G SNP Effect on Striatal Dopamine Response to an IV Opiate
Brief Title: Genetic Effects on Dopamine Response to an Opiate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 130061; 13-AA-0061
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Polymorphism-Genetic; Pain; Addiction
Keywords: Opiate Receptor; Genotype; PET Imaging
MeSH Terms: conditions — Pain; Behavior, Addictive | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Crossover study - participants receive active and placebo treatments in randomized order.
Who Masked: Participant, Investigator
Masking Description: Bliniding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Morphine (Experimental): Morphine injection 10 mg/70kg
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Saline injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine
  Arms: Morphine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background:

- Small differences in genes may alter responses to drugs. One gene that has different forms is the mu opioid receptor gene. People with one form of this gene are more sensitive to alcohol. People with a different form are sometimes more sensitive to pain. Morphine and other prescription pain pills produce pain relief by acting at the mu opioid receptor. Researchers want to see the effect of morphine on brain reward and subjective effects. Morphine is a strong but short-acting pain medication that is sometimes used for anesthesia during surgery.

Objectives:

- To compare the effect of morphine on brain measures of dopamine release using imaging.

Eligibility:

- Individuals between 21 and 55 years of age who have previously taken pain pills prescribed to treat pain from a medical or dental procedure.

Design:

* This study has a screening phase and a study phase. The screening phase involves one or two visits of 5 to 6 hours. The study phase consists of 4 study visits. Each study visit will take about 8 hours.
* Participants will be screened with a medical and psychiatric history and physical exam. They will be asked about drinking and drug-taking history, and any family history of alcoholism or drug abuse. Blood, urine, and breath samples will be collected.
* During the first study visit, an MRI scan may be performed, questionnaires completed, and a blood sample collected for genetic testing.
* During study visit 2, participants will test their pain sensitivity by placing one hand in cold water. Pupil diameter will be measured after the sensitivity test. After a blood sample is taken, participants will receive the morphine or a salt solution. The sensitivity test and pupil diameter test will be repeated. Final blood samples will be collected. A brief physical exam will also be performed.
* During study visits 3 and 4, participants will receive morphine or a salt solution during a PET scan. Questionnaires to assess subjective effects will be administered. Final blood samples will be collected. A brief physical exam will also be performed.
* Participants will stay in the clinic until the effects of the drug have worn off after study visits 2, 3, and 4.
* About 1 week after the study session, participants will have a follow-up phone call.

DETAILED DESCRIPTION:
Objectives

Mesolimbic dopamine (DA) release is a key signal for drug reward, and endogenous opioids are thought to exert their effects in part by modulating the activity of this system. A functional µ-opioid receptor (OPRM1) A118G single nucleotide polymorphism (SNP) has been associated with increased risk for heroin addiction in some studies. This polymorphism has been shown to confer differential pain sensitivity and to alter the release of DA following an alcohol challenge. The objective of this study is to examine the role of the A118G OPRM1 polymorphism for responses to a challenge of an opiate (morphine) with regard to psycho-physiological variables measured in the laboratory and for brain dopamine release measured by [11C]raclopride PET.

Study Population

Healthy male participants who have had experience with oral prescription analgesics (e.g., Oxycontin, Vicodin, Percocet, oxycodone) will be recruited for the study. These volunteers will be screened to obtain samples of two groups of subjects: 1) persons homozygous for the major 118A allele (118AA genotype); 2) persons carrying one or two copies of the variant 118G allele (118AG or 118GG genotype, hereafter called 118GX). We will recruit up to 120 participants to obtain 40 completers per genotype for the study.

Design

We will compare the response of these groups to a challenge with morphine given intravenously. Participants will receive a standardized IV challenge of morphine (10.0 mg/70 kg over 1 minute; morphine concentration 2 mg/ml). Pre and post injection measures will be made in two areas: 1) subjective response as measured by standardized questionnaires, and 2) measures of physiological response, including pupil response to light, respiratory rate, oxygen saturation and a pain rating from putting a hand in cold water and blood chemistries. In addition, during this visit, participants will wear the AutoSense mobile physiological monitor; parameters measured by AutoSense include respiration rate, heart rate, heart-rate variability, skin conductance, and activity level. The injection will be repeated in all participants in the PET scanner, once with morphine and once with normal saline. Dopamine release will be assessed by determining the difference between the binding potential for [11C]raclopride, a positron emitter labeled ligand which binds preferentially to D2 receptors during saline administration and its binding potential during morphine administration.

Outcome measures

We hypothesize that 118GX subjects will have significantly different subjective response to the challenge than 118AA subjects as observed in participants receiving alcohol in a similar study (Ramchandani et al. 2011). However, the genotype effect on the response may be opposite from the effect of genotype on the alcohol response. We also hypothesize that the PET studies with [11C]raclopride will show that 118GX subjects have less dopamine release during morphine administration than 118 AA subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male participants between 21-55 years of age.
  2. Good health as determined by medical history, physical exam, EKG and lab tests.
  3. Current non-smokers or light smokers or e-cigarette users (<20 cig/week) who can easily abstain from smoking or using e-cigarettes for 1-2 days/week.
  4. Current non-drinkers or social drinkers who do not meet past or current DSM IV criteria for alcohol abuse or alcohol dependence.
  5. An equal number of final participants will be of OPRM1 118 A/A vs. 118A/G or 118G/G genotype. This means that after the first group (n40) is complete then only participants with the required genotype for the other group will be included.
  6. Prior opiate use, at least one experience with one of the opiates listed in Appendix 1 of the protocol.
  7. Comprehension/fluency with English Language.

EXCLUSION CRITERIA:<TAB>

1. Current or prior history of any significant disease, including cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, or a positive hepatitis or HIV test at screening, disorders that could make administration of an opiate more risky (e.g., asthma, COPD, sleep apnea, or other breathing disorders; liver or kidney disease; thyroid disorder; trouble swallowing, or a blockage in the digestive tract (stomach or intestines); neurologic disorders (e.g., a history of head injury or brain tumor, epilepsy or other seizure disorder, CVA, migraine in treatment, etc.); low blood pressure; hypertension; neuromuscular disorder; gallbladder disease; Addison's disease or other adrenal gland disorders; enlarged prostate, urination problems)
2. Current Axis-I psychiatric illness as determined by the Structured Clinical Interview for DSM IV disorders (SCID).
3. Current or prior history of any alcohol or drug dependence as determined by the Structured Clinical Interview for DSM IV disorders (SCID).
4. Positive result on urine screen for illicit drugs.
5. Medication Use:

   1. Current chronic prescription or over the counter medications or use of prescription or OTC medications known to interact with dopamine receptors within 2 weeks of the study
   2. Drugs known to inhibit or induce enzymes that metabolize opiates should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram.
   3. Cough-and-cold preparations that contain anti-histamines or opiate pain medicines will be withheld for at least 72 hours prior to each study session.
   4. Drugs that may interfere with the BOLD MRI signal within 2 weeks of the study. These include, but may not be limited to: muscle relaxants or respiratory, cardiovascular or anticonvulsant medications
6. Morbid obesity (BMI >40 kg/m2)
7. Previous negative effects of opioid administration
8. Presence of certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia. Justification: Implanted devices may increase the risk of MRI scanning and/or adversely affect the quality of the data; body morphology may prevent optimal positioning in the scanner and thus affect the quality of the data; participants with claustrophobia may find the MRI scan too unpleasant and may exhibit excess movement that will adversely affect the quality of the data. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Questions concerning suitability for scanning will be referred to the Medical Advisory Investigator. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their first visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner.
9. Conditions restricting participant's ability to lie flat for up to two hours (such as coagulopathies, superficial or deep vein thrombosis, or musculoskeletal abnormalities). Justification: PET scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g., chronic back pain, significant scoliosis) or dangerous (e.g., familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort.
10. Head trauma leading to loss of consciousness for more than 5 min or hospitalization
11. Exposure to ionizing radiation from research studies that, in combination with the study tracer, would result in cumulative exposure of >5 rem within the previous 12 month period
12. Self-reported and/or observed signs, symptoms, or diagnosis of Raynaud's or Buerger's disease (e.g., pain in hands or feet at times of rest, during/following cold exposure or stress, any significant color changes in hands or toes). Additionally, medical staff will be present to watch for these symptoms during the actual cold pressor test.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06-13; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The protocol does not outline a plan for data sharing. Samples and data will be transferred to a repository for analysis of exploratory outcomes beyond the primary objectives of the study, after IRB approval.

REFERENCES:
- [Background] Barr CS, Schwandt M, Lindell SG, Chen SA, Goldman D, Suomi SJ, Higley JD, Heilig M. Association of a functional polymorphism in the mu-opioid receptor gene with alcohol response and consumption in male rhesus macaques. Arch Gen Psychiatry. 2007 Mar;64(3):369-76. doi: 10.1001/archpsyc.64.3.369. PMID 17339526
- [Background] Bart G, Heilig M, LaForge KS, Pollak L, Leal SM, Ott J, Kreek MJ. Substantial attributable risk related to a functional mu-opioid receptor gene polymorphism in association with heroin addiction in central Sweden. Mol Psychiatry. 2004 Jun;9(6):547-9. doi: 10.1038/sj.mp.4001504. No abstract available. PMID 15037869
- [Background] Callaghan RC, Cunningham JK, Verdichevski M, Sykes J, Jaffer SR, Kish SJ. All-cause mortality among individuals with disorders related to the use of methamphetamine: a comparative cohort study. Drug Alcohol Depend. 2012 Oct 1;125(3):290-4. doi: 10.1016/j.drugalcdep.2012.03.004. Epub 2012 Apr 13. PMID 22503689
- [Derived] Spagnolo PA, Kimes A, Schwandt ML, Shokri-Kojori E, Thada S, Phillips KA, Diazgranados N, Preston KL, Herscovitch P, Tomasi D, Ramchandani VA, Heilig M. Striatal Dopamine Release in Response to Morphine: A [11C]Raclopride Positron Emission Tomography Study in Healthy Men. Biol Psychiatry. 2019 Sep 1;86(5):356-364. doi: 10.1016/j.biopsych.2019.03.965. Epub 2019 Mar 15. PMID 31097294
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-AA-0061.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects were consented for the trial, but 10 subjects were found eligible to start the study.
Groups:
- First Morphine, Then Placebo; First Placebo, Then Morphine: All participants received in counterbalanced order an IV infusion of morphine (10 mg/70 kg) or an equivalent volume of normal saline over 20-30 s
Period: Study Session 1
Arm/Group | First Morphine, Then Placebo | First Placebo, Then Morphine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Study Session 2
Arm/Group | First Morphine, Then Placebo | First Placebo, Then Morphine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants who started the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 11C Raclopride Binding Potential in Caudate
Description: Binding potential measured using regions-of-interest analysis of PET data. Parametric Binding Potential (BPND) images were obtained using the Simple Reference Tissue Model 2 (SRTM2), with cerebellum as the reference region. BPND is computed in units of mCi/ml reflecting the radioactivity (milliCuries or mCi) per unit volume (milliliters or ml) in specific brain regions. Reduction in raclopride binding is attributed to competition with endogenous dopamine, and has been shown to be proportional to the magnitude of Dopamine (DA) release.
Time Frame: 90 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: mCi/ml
Groups:
- Morphine; Placebo: All participants received in counterbalanced order an IV infusion of morphine (10 mg/70 kg) or an equivalent volume of normal saline (placebo) over 20-30 s
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
mCi/ml | 3.25 (0.4) | 3.45 (0.5)

2. Primary Outcome: 11C Raclopride Binding Potential in Nucleus Accumbens
Description: as for outcome 1
Time Frame: 90 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: mCi/ml
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
mCi/ml | 2.68 (0.5) | 2.84 (0.4)

3. Primary Outcome: 11C Raclopride Binding Potential in Putamen
Description: as for outcome 1
Time Frame: 90 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: mCi/ml
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
mCi/ml | 3.9 (0.4) | 4.11 (0.6)

4. Primary Outcome: 11C Raclopride Binding Potential in Ventral Pallidum
Description: as for outcome 1
Time Frame: 90 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: mCi/ml
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
mCi/ml | 2.68 (0.4) | 2.94 (0.5)

5. Secondary Outcome: Subjective Perception of Morphine Effect - Feel Drug
Description: Area under the curve of the subjective perception-time course - Feel Drug. Subjective responses as measured by the Drug Effects Questionnaire [DEQ]. The DEQ consists of simple, face-valid, visual analog scale (VAS) questions on which people report their subjective states after ingesting a substance. The analog scale of responses ranges from "not at all" to "extremely", and the numeric scale ranges from 0 to 100. Due to skewness of individual time points; areas under the curve (AUC) for these ratings across individual time points (0, 10, 20, 30, 40, 50 and 60 min) were compared. AUC is computed using the trapezoidal rule and has a range of values from 0 to 5500, where 0 reflects no subjective perception at any time point and 5500 reflects maximal subjective perception (score of 100) at all time points after drug administration.
Time Frame: 60 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: Units on a scale * min
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale * min | 3942.8 (856.1) | 176 (553.1)

6. Secondary Outcome: Subjective Perception of Morphine Effect - Feel High
Description: Area under the curve of the subjective perception-time course - Feel High. Subjective responses as measured by the Drug Effects Questionnaire [DEQ]. The DEQ consists of simple, face-valid, visual analog scale (VAS) questions on which people report their subjective states after ingesting a substance. The analog scale of responses ranges from "not at all" to "extremely", and the numeric scale ranges from 0 to 100. Due to skewness of individual time points; areas under the curve (AUC) for these ratings across individual time points (0, 10, 20, 30, 40, 50 and 60 min) were compared. AUC is computed using the trapezoidal rule and has a range of values from 0 to 5500, where 0 reflects no subjective perception at any time point and 5500 reflects maximal subjective perception (score of 100) at all time points after drug administration.
Time Frame: 60 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: Units on a scale * min
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale * min | 3729.4 (1132.1) | 175 (553.4)

7. Secondary Outcome: Subjective Perception of Morphine Effect - Like Drug
Description: Area under the curve of the subjective perception-time course - Like Drug. Subjective responses as measured by the Drug Effects Questionnaire [DEQ]. The DEQ consists of simple, face-valid, visual analog scale (VAS) questions on which people report their subjective states after ingesting a substance. The analog scale of responses ranges from "not at all" to "extremely", and the numeric scale ranges from 0 to 100. Due to skewness of individual time points; areas under the curve (AUC) for these ratings across individual time points (0, 10, 20, 30, 40, 50 and 60 min) were compared. AUC is computed using the trapezoidal rule and has a range of values from 0 to 5500, where 0 reflects no subjective perception at any time point and 5500 reflects maximal subjective perception (score of 100) at all time points after drug administration.
Time Frame: 60 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: Units on a scale * min
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale * min | 3078.9 (1881.14) | 2628.5 (952.1)

8. Secondary Outcome: Subjective Perception of Morphine Effect - Want More
Description: Area under the curve of the subjective perception-time course - Want More. Subjective responses as measured by the Drug Effects Questionnaire [DEQ]. The DEQ consists of simple, face-valid, visual analog scale (VAS) questions on which people report their subjective states after ingesting a substance. The analog scale of responses ranges from "not at all" to "extremely", and the numeric scale ranges from 0 to 100. Due to skewness of individual time points; areas under the curve (AUC) for these ratings across individual time points (0, 10, 20, 30, 40, 50 and 60 min) were compared. AUC is computed using the trapezoidal rule and has a range of values from 0 to 5500, where 0 reflects no subjective perception at any time point and 5500 reflects maximal subjective perception (score of 100) at all time points after drug administration.
Time Frame: 60 minutes following injection
Population: The analyses included only those subjects who completed both PET sessions (active and placebo)
Measure: Mean (Standard Deviation); unit: Units on a scale * min
Arm/Group | Morphine | Placebo
Number analyzed (Participants) | 10 | 10
Units on a scale * min | 1601.1 (1352.4) | 1277 (1674.6)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Morphine; Placebo: All participants received in counterbalanced order an IV infusion of morphine (10 mg/70 kg) or an equivalent volume of normal saline over 20-30 s
Arm/Group | Morphine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=10) | Placebo (N=10)
Dizziness (Cardiac disorders) | 4 | 0
dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Sedation (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT01878006/Prot_SAP_000.pdf